CLINICAL TRIAL: NCT03012906
Title: Prospective Multicenter Registry of the Combination of Antiplatelet Agents and Anticoagulant in Atrial Fibrillation Patients With a CHA2DS2VASc Score >1 Undergoing Percutaneous Coronary Interventions
Brief Title: Registry of the Combination of Antiplatelet Agents and Anticoagulant in Atrial Fibrillation Patients With a CHA2DS2VASc Score >1 Undergoing Percutaneous Coronary Interventions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-16
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: the prevalence of ischemic events

SUMMARY:
Patients undergoing percutaneous coronary intervention (PCI) with stent implantation and requiring chronic anticoagulation for atrial fibrillation (AF) with a CHA2DS2-VASc >1 are required to receive triple antithrombotic therapy . This triple therapy includes dual antiplatelet therapy with clopidogrel and aspirin in combination with an oral anticoagulant with either a vitamin K antagonist (VKA) or an oral anticoagulant (NOAC).

Recently NOAC, inhibiting the IIa (dabigatran) or Xa (rivaroxaban and apixaban) in the coagulation cascade have demonstrated non inferiority compared to VKA to prevent thrombo-embolic events in non-valvular AF for patients with a CHA2DS2-VASc >1 . Interestingly, NOAC are associated with a reduced fatal bleeding rate compared to VKA. Overall they seem to result in a lower bleeding rate compared to VKA in association with antiplatelet agents.

Recently European guidelines regarding patients requiring chronic anticoagulant therapy and undergoing coronary stent implantation have been updated. However they are based on an expert consensus because of the scarce data available.

These guidelines advocate the combination of dual antiplatelet therapy with clopidogrel and aspirin in combination with the lower dose of OAC or VKA with a target INR between 2 and 2.5 . The triple therapy should be prescribed for 1 to 6 months depending on the bleeding and thrombotic risk and the clinical setting. In patients with high bleeding risk the guidelines suggest that a sole antiplatelet agent could be used in addition to anticoagulation following the WOEST study . In the recently published ESC guidelines on the management of atrial fibrillation, despite the lack of new data, the expert advocate triple therapy followed by dual antiplatelet therapy in most patients for 12 months.

The recently published PIONEER study reinforced the possibility of the use of rivaroxaban in these patients. In this trial including ACS and not ACS patients undergoing PCI rivaroxaban 15 mg in addition to a P2Y12 ADP receptor antagonist was associated with less clinically relevant bleeding compared to triple therapy with VKA- aspirin and clopidogrel and similar efficacy .

ELIGIBILITY:
Inclusion Criteria:

1. age over 18 years old
2. signed informed consent
3. requiring PCI (with stent placement) with subsequent need for antiplatelet therapy
4. FA requiring chronic anticoagulation (CHA2DS2-VASc >1, except women with a score =1).

Exclusion Criteria:

1. pregnancy or lactation
2. age <18 or not able to give an informed consent
3. no informed consent
4. no health insurance
5. prisoners
6. contra indication to antiplatelet therapy
7. intra cardiac thrombus
8. active bleeding Known bleeding diathesis (i.e. history of ICH, GI bleeding)
9. severe kidney failure (eGFR < 30 mL/min/1.73 m²)
10. severe hepatic failure (Child-Pugh class B or C)
11. contra indication to OAC or VKA
12. hypertrophic myocardiopathy
13. valvular prosthesis
14. history of peptic ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing percutaneous coronary intervention (PCI)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Number of deaths | 2 years
Number of myocardial infarctions | 2 years
Number of strokes | 2 years

SECONDARY OUTCOMES:
The prevalence of bleeding events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille; Laurent bonello, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No